CLINICAL TRIAL: NCT03220204
Title: A Positive Psychology Intervention to Promote Health Behaviors in Heart Failure: a Randomized, Controlled Pilot Trial
Brief Title: Researching Emotions And Cardiac Health: Phase III
Acronym: REACH III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christopher Celano, Assistant Psychiatrist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5K23HL123607-03 (NIH); 5K23HL123607-03 (NIH)
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Results first posted 2020-04-03 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Congestive Heart Failure; Emotions; Patient Compliance
Keywords: Heart Failure; Positive Psychology; Adherence to Health Behaviors
MeSH Terms: conditions — Heart Failure; Patient Compliance

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded, controlled trial
Who Masked: Outcomes Assessor
Masking Description: Participants and treating study staff will be aware of the participant's treatment condition. However, follow-up assessments will be performed by a study staff member that is masked to the participant's treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PP-based health behavior intervention (Experimental): Participants will undergo a 12-week, Positive Psychology (PP)-based health behavior intervention. Each weekly session will include (a) a review of the week's PP exercise, (b) a discussion of the rationale of the next week's PP exercise through a guided review of the PP manual, and (c) assignment of the next week's PP exercise. Additionally for the goal-setting portion, participants will (a) review their goals and behaviors from the prior week, (b) discuss techniques for improving health behavior adherence (e.g., monitoring physical activity, reading nutrition labels), and (c) set goals for the next week.
  Interventions: Behavioral: PP-based health behavior intervention
- MI-based educational control condition (Experimental): Participants will undergo 12 weekly phone sessions to learn about a different health behavior topic related to cardiac health. This Motivational Interviewing (MI)-based educational control condition will introduce these participants to motivational interviewing topics in concert with the health behavior education topics.
  Interventions: Behavioral: MI-based educational control condition
- Treatment as Usual (TAU) (No Intervention): Participants in the Treatment as Usual (TAU) group will not receive any interventions between the baseline visit and follow-up visits.

INTERVENTIONS:
Behavioral: PP-based health behavior intervention — The positive psychology exercises include 3 modules: gratitude-based activities, strength-based activities, and meaning-based activities. The goal-setting portion of the program focuses primarily on physical activity (8 weeks) but also includes 4 weeks focusing on diet and medication adherence.
  Arms: PP-based health behavior intervention
Behavioral: MI-based educational control condition — The MI-based educational program includes information on five topics: (1) information about heart disease and risk factors for worsening heart disease, (2) physical activity, (3) a heart-healthy diet, (4) medication adherence, and (5) stress management.
  Arms: MI-based educational control condition

SUMMARY:
The focus of this study is to examine the feasibility, acceptability, and preliminary impact of a 12-week, telephone-delivered, positive psychology (PP)-based health behavior intervention in a group of patients with mild to moderate heart failure (HF), compared to a motivational interviewing- (MI-) based education condition and treatment as usual (TAU).

DETAILED DESCRIPTION:
The investigators are proposing a study that will focus on the implementation of a novel PP-based health behavior intervention that is adapted for patients with HF. The MGH inpatient units, MGH Heart Center, and MGH primary care clinic outpatients will serve as the source of participants for the study, with patients who have a diagnosis of HF serving as potential participants. The investigators will enroll 60 HF patients, who will take part in a 12-week PP-based health behavior intervention.

In this project, the investigators hope to do the following:

1. Test a 12-week, telephone-delivered health behavior intervention utilizing PP exercises and systematic goal-setting in a three-arm, randomized, controlled pilot trial in patients with mild to moderate HF (N=60).
2. Determine whether this optimized intervention is feasible in a small cohort of HF patients.
3. Explore potential benefits of the intervention on outcomes of interest (e.g., psychological health, functioning, and health behavior adherence) compared to a motivational interviewing- (MI) based education condition and treatment as usual (TAU).

Baseline information about enrolled participants will be obtained from the patients, care providers, and the electronic medical record as required for characterization of our population. This information will include data regarding medical history (history of prior acute coronary syndrome, coronary artery disease, coronary artery bypass graft, congestive HF, hypertension, diabetes mellitus, hyperlipidemia, and current smoking), current medical variables (renal function, left ventricular ejection fraction, NYHA class), medications, and sociodemographic data (age, gender, race/ethnicity, living alone).

Participants will undergo two in person visits during which they will meet with study staff in person (or if preferred over the phone). In their first visit, they will answer questionnaires related to psychological and physical health and functioning and will be asked to wear an accelerometer for one week to measure their baseline physical activity. At their second in-person visit, they will be randomized to receive (1) the PP-based health behavior intervention, (2) the MI-based educational condition, or (3) TAU. Participants in the TAU group will not receive any additional intervention but will complete follow-up phone calls at 12 and 24 weeks.

Following randomization, participants in the two treatment groups will be provided a treatment manual corresponding with their treatment condition with weekly exercises, along with a copy of the Learning to Live with Heart Failure guide. The appropriate intervention will be introduced, and the first exercise will be assigned. Finally, participants in both treatment groups will receive a personal step counter to use over the course of the study.

Following the second in-person visit, participants in the PP-based intervention and MI-based control condition groups will complete twelve 30- to 45-minute weekly phone sessions with a study trainer. The phone sessions primarily will include a review of the prior week's session content and a discussion of the rationale and assignment of the next week's exercise/assignment.

At Weeks 12 and 24, a member of the study staff will call participants to repeat the self-report questionnaires that were administered at baseline. At these two time points, participants also will be asked to wear an accelerometer for an additional 7 days to measure physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with NYHA class I, II, or III HF admitted to an MGH inpatient unit or outpatients at the MGH Heart Center or MGH-affiliated primary care clinic. Patients with NYHA class IV HF have ongoing HF symptoms at rest, making it difficult for them to increase physical activity and other health behaviors; therefore, they will not be included. HF diagnosis will be confirmed via chart review and with the patient's treatment team as needed.
* Suboptimal adherence to health behaviors. This will be defined as a total score of ≤15 on three Medical Outcomes Study Specific Adherence Scale (MOS) items regarding diet/exercise/medications. The MOS has been used in multiple prior studies assessing adherence in cardiac patients, including our own studies in this population. This threshold score on the MOS will ensure that all participants will have the potential to improve their health behaviors.

Exclusion Criteria:

* Cognitive deficits impeding a participant's ability to provide informed consent or participate, assessed via a 6-item cognitive test that is sensitive and specific for screening for cognitive impairment in research participants.
* Medical conditions precluding interviews or likely to lead to death within 6 months.
* Inability to speak English, inability to read or write, inability to walk, or lack of a telephone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Celano, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Celano CM, Freedman ME, Harnedy LE, Park ER, Januzzi JL, Healy BC, Huffman JC. Feasibility and preliminary efficacy of a positive psychology-based intervention to promote health behaviors in heart failure: The REACH for Health study. J Psychosom Res. 2020 Dec;139:110285. doi: 10.1016/j.jpsychores.2020.110285. Epub 2020 Oct 29. PMID 33160091

RESULTS

PARTICIPANT FLOW:
Groups:
- MI-based Educational Control Condition: Participants will undergo 12 weekly phone sessions to learn about a different health behavior topic related to cardiac health. They will also be introduced to motivational interviewing topics in concert with the health behavior education topics.
  Motivational Interviewing (MI)-based educational control condition: The MI-based educational program includes information on five topics: (1) information about heart disease and risk factors for worsening heart disease, (2) physical activity, (3) a heart-healthy diet, (4) medication adherence, and (5) stress management.
Period: Overall Study
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU)
Started | 15 | 15 | 15
Completed | 14 | 13 | 12
Not Completed | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Population: While 50 participants enrolled in this study, only 45 participants were randomized to a condition as 2 participants withdrew consent, 1 participant terminated consent, 1 participant was lost to follow-up, and 1 participant did not provide the data necessary to be randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (8.5) | 74.6 (10.4) | 71.8 (10.6) | 70.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 4 | 12
  Male | 13 | 9 | 11 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 15 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 4
  White | 13 | 12 | 14 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 45
Positive and Negative Affect Schedule (PANAS) [Mean (Standard Deviation); unit: units on a scale] — The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with HF, will be used to measure positive affect (Range: 10-50). Higher scores indicate higher levels of positive affect.
  units on a scale | 31.53 (7.95) | 33.93 (7.21) | 32.33 (5.81) | 32.60 (6.96)
Life Orientation Test-Revised (LOT-R) [Mean (Standard Deviation); unit: units on a scale] — Life Orientation Test-Revised (LOT-R) is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Higher scores indicate higher levels of dispositional optimism.
  units on a scale | 17.33 (3.64) | 18.13 (4.55) | 15.73 (4.77) | 17.07 (4.37)
State Optimism Measure (SOM) [Mean (Standard Deviation); unit: units on a scale] — The State Optimism Measure (SOM) will be used to measure state optimism (Range: 7-35). Higher scores indicate higher levels of state optimism.
  units on a scale | 26.33 (4.85) | 26.93 (5.54) | 27.67 (4.51) | 26.98 (4.90)
Hospital Anxiety and Depression Scale (HADS) anxiety subscale [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale (HADS)-anxiety subscale was be used to measure anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21).
  units on a scale | 6.47 (3.72) | 6.33 (4.01) | 5.60 (4.56) | 6.13 (4.04)
Hospital Anxiety and Depression Scale (HADS) depression subscale [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale (HADS)-depression subscale was be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of depression.
  units on a scale | 5.07 (3.35) | 5.40 (3.92) | 5.13 (4.02) | 5.20 (3.69)
Kansas City Cardiomyopathy Questionnaire (KCCQ) [Mean (Standard Deviation); unit: units on a scale] — The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a well-validated questionnaire of health status in HF. The full scale will be used to measure HF-specific health-related QoL (HRQoL), and an eight-question subset of the KCCQ will be used as a measure of HF symptoms (QoL score range: 0-100; total symptom score range: 0-100). Higher QoL scores indicate better HF specific health-related QoL, and higher total symptom scores indicate fewer symptoms.
  units on a scale | 75.36 (19.16) | 68.91 (24.35) | 78.15 (14.99) | 74.14 (19.81)
Medical Outcomes Study Short Form-12 (SF-12) [Mean (Standard Deviation); unit: units on a scale] — The Medical Outcomes Study Short Form-12 (SF-12) will be used to measure quality of life. This is an instrument which has been used in multiple cardiac studies in the past (SF-12 Mental Composite Score and Physical Composite Score Range: 0-100 each). Higher scores indicate higher level of health related QoL.
  units on a scale
    Physical Health Composite Score | 42.13 (10.05) | 37.94 (13.68) | 40.14 (10.40) | 40.07 (11.36)
    Mental Health Composite Score | 42.21 (11.20) | 50.26 (8.72) | 48.22 (9.99) | 46.90 (10.38)
Medical Outcomes Study Specific Adherence Scale (MOS SAS) [Mean (Standard Deviation); unit: units on a scale] — Three Medical Outcomes Study Specific Adherence Scale (MOS SAS) items assessing medication, diet, and exercise, will be measured individually and as a composite score (Range: 3-18). Higher scores indicate better adherence to health behaviors.
  units on a scale | 11.87 (2.33) | 12.60 (2.10) | 12.73 (1.28) | 12.40 (1.95)
Scored Sodium Questionnaire (SSQ) [Mean (Standard Deviation); unit: units on a scale] — The Scored Sodium Questionnaire (SSQ) is a self-report scale that assesses the frequency with which participants consume a variety of sodium-containing foods, ranging from "Rarely or Never Eaten" to "At Least Once Daily." It is used to calculate daily sodium intake (Range: 0-215). Higher scores indicate higher sodium intake.
  units on a scale | 71.10 (29.09) | 64.90 (27.79) | 64.37 (21.15) | 66.79 (25.82)
Self-Reported Medication Adherence (SRMA) [Mean (Standard Deviation); unit: percentage] — The Self-Reported Medication Adherence (SRMA) asks what percent of the time (in 10% increments) participants took all of their medications as prescribed in the past week and in the past 2 weeks (Range: 0-100).
  percentage | 95.33 (5.16) | 96.67 (4.88) | 96.67 (6.17) | 96.22 (5.35)
Physical Activity [Mean (Standard Deviation); unit: steps/day] — Assessed by ActiGraph GT3X+ step counters which are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. We will measure both number of steps per day (primary physical health outcome).
  steps/day | 3465 (1484) | 3458 (1616) | 4195 (2375) | 3706 (1857)
Moderate to Vigorous Physical Activity [Mean (Standard Deviation); unit: minutes/day] — Assessed with ActiGraph GT3X+ step counters, which are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness.
  minutes/day | 7.5 (6.8) | 5.9 (6.9) | 15.2 (19.8) | 9.5 (13.1)
Feasibility of Actigraph [Count of Participants; unit: Participants] — Feasibility will be measured by examining the number of participants who provide adequate Actigraph data, defined in this study as at least 480 minutes for 5 days.
  Participants | 15 | 15 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the PP-based Health Behavior Intervention
Description: Feasibility will be measured by examining the number of completed exercises for individuals randomized to the Positive Psychology (PP)-based intervention.
Time Frame: Change between baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: sessions completed out of 12 sessions
Groups:
- PP-based Health Behavior Intervention: Participants will undergo a 12-week, PP-based health behavior intervention. Each weekly session will include (a) a review of the week's PP exercise, (b) a discussion of the rationale of the next week's PP exercise through a guided review of the PP manual, and (c) assignment of the next week's PP exercise. Additionally for the goal-setting portion, participants will (a) review their goals and behaviors from the prior week, (b) discuss techniques for improving health behavior adherence (e.g., monitoring physical activity, reading nutrition labels), and (c) set goals for the next week.
  PP-based health behavior intervention: The positive psychology exercises include 3 modules: gratitude-based activities, strength-based activities, and meaning-based activities. The goal-setting portion of the program focuses primarily on physical activity (8 weeks) but also includes 4 weeks focusing on diet and medication adherence.
Arm/Group | PP-based Health Behavior Intervention
Number analyzed (Participants) | 15
sessions completed out of 12 sessions | 8.7 (4.9)

2. Secondary Outcome: Acceptability of the Exercises
Description: Participants receiving the PP-based health behavior intervention will provide ratings of ease and utility after each exercise, measured on a 10-point Likert scale.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: rating out of 10
Arm/Group | PP-based Health Behavior Intervention
Number analyzed (Participants) | 15
rating out of 10
  Ease | 7.5 (1.7)
  Utility | 7.5 (1.6)

3. Secondary Outcome: Immediate Impact of the Exercises
Description: Participants receiving the PP-based health behavior intervention will provide ratings of optimism and positive affect, before and after each exercise, measured on a 10-point Likert scale.
Time Frame: Weekly, up to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-based Health Behavior Intervention
Number analyzed (Participants) | 15
units on a scale
  Optimism | 0.64 (1.14)
  Positive Affect | 0.97 (1.38)

4. Secondary Outcome: Change in PANAS Scores (Primary Psychological Outcome)
Description: The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with HF, will be used to measure positive affect (Range: 10-50). Change was calculated by subtracting the score at baseline from the score at 12 and 24 weeks. Higher scores indicate higher levels of positive affect.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: Not all participants provided follow-up data at both timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU)
Number analyzed (Participants) | 14 | 14 | 14
units on a scale
  12 weeks | 5.38 (7.84) | 2.50 (8.26) | 2.50 (5.60)
  24 weeks: number analyzed (Participants) | 14 | 13 | 12
  24 weeks | 5.43 (5.15) | -0.46 (7.29) | 3.75 (7.44)

5. Secondary Outcome: Changes in LOT-R Scores
Description: Life Orientation Test-Revised (LOT-R) is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Change was calculated by subtracting the score at baseline from the score at 12 and 24 weeks. Higher scores indicate higher levels of dispositional optimism.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: Not all participants provided follow-up data at both timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- MI-based Educational Control Condition: Participants will undergo 12 weekly phone sessions to learn about a different health behavior topic related to cardiac health. They will also be introduced to motivational interviewing topics in concert with the health behavior education topics.
  MI-based educational control condition: The MI-based educational program includes information on five topics: (1) information about heart disease and risk factors for worsening heart disease, (2) physical activity, (3) a heart-healthy diet, (4) medication adherence, and (5) stress management.
- Treatment as Usual (TAU): Participants in the TAU group will not receive any interventions between the baseline visit and follow-up visits.
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU)
Number analyzed (Participants) | 14 | 14 | 14
units on a scale
  12 weeks | 2.43 (4.18) | 1.29 (3.05) | 2.93 (5.92)
  24 weeks: number analyzed (Participants) | 14 | 13 | 12
  24 weeks | 3.50 (3.35) | 1.23 (4.66) | 2.83 (6.62)

6. Secondary Outcome: Changes in SOM Scores
Description: The State Optimism Measure (SOM) will be used to measure state optimism (Range: 7-35). Change was calculated by subtracting the score at baseline from the score at 12 and 24 weeks. Higher scores indicate higher levels of state optimism.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: Not all participants provided follow-up data at both timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU)
Number analyzed (Participants) | 14 | 14 | 14
units on a scale
  12 weeks | 2.14 (4.38) | 1.29 (4.63) | 2.36 (3.97)
  24 weeks: number analyzed (Participants) | 14 | 13 | 12
  24 weeks | 2.00 (4.61) | 1.38 (5.74) | -0.17 (5.61)

7. Secondary Outcome: Changes in HADS-Anxiety Subscale Scores
Description: The Hospital Anxiety and Depression Scale (HADS)-anxiety subscale was be used to measure anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Change was calculated by subtracting the score at baseline from the score at 12 weeks and 24 weeks. Higher scores indicate higher levels of anxiety.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: Not all participants provided follow-up data at both timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU)
Number analyzed (Participants) | 14 | 14 | 14
units on a scale
  12 weeks | -1.79 (3.42) | -2.00 (2.54) | -2.07 (3.85)
  24 weeks: number analyzed (Participants) | 14 | 13 | 12
  24 weeks | -2.21 (1.72) | -1.69 (3.47) | -2.50 (4.44)

8. Secondary Outcome: Change in HADS-Depression Subscale Scores
Description: The Hospital Anxiety and Depression Scale (HADS)-depression subscale was be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Change was calculated by subtracting the score at baseline from the score at 12 weeks and 24 weeks. Higher scores indicate higher levels of depression.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: Not all participants provided follow-up data at both timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU)
Number analyzed (Participants) | 14 | 14 | 14
units on a scale
  12 weeks | -1.57 (2.47) | -0.93 (2.53) | -1.00 (2.63)
  24 weeks: number analyzed (Participants) | 14 | 13 | 12
  24 weeks | -1.57 (2.24) | -0.38 (5.12) | -1.00 (3.33)

9. Secondary Outcome: Changes in KCCQ Scores (Primary Functional Outcome)
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a well-validated questionnaire of health status in HF. The full scale will be used to measure HF-specific health-related QoL (HRQoL), and an eight-question subset of the KCCQ will be used as a measure of HF symptoms (QoL score range: 0-100; total symptom score range: 0-100). Change was calculated by subtracting the score at baseline from the score at 12 weeks and 24 weeks. Higher QoL scores indicate better HF specific health-related QoL, and higher total symptom scores indicate fewer symptoms.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: Not all participants provided follow-up data at both timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU)
Number analyzed (Participants) | 14 | 14 | 14
units on a scale
  12 weeks HRQoL | 7.74 (24.99) | 4.76 (23.28) | 10.12 (13.94)
  12 weeks Total Symptom | 2.31 (21.39) | -1.19 (10.89) | 2.60 (16.65)
  24 weeks HRQoL: number analyzed (Participants) | 14 | 13 | 12
  24 weeks HRQoL | 1.19 (22.13) | 7.05 (26.75) | 10.42 (12.87)
  24 weeks Total Symptom: number analyzed (Participants) | 14 | 13 | 12
  24 weeks Total Symptom | 1.93 (18.49) | -5.37 (14.14) | 0.87 (16.66)

10. Secondary Outcome: Changes in SF-12 Scores
Description: The Medical Outcomes Study Short Form-12 (SF-12) will be used to measure quality of life. This is an instrument which has been used in multiple cardiac studies in the past (SF-12 Mental Composite Score and Physical Composite Score Range: 0-100 each). Change was calculated by subtracting the score at baseline from the score at 12 weeks and 24 weeks. Higher scores indicate higher level of health related QoL.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: Not all participants provided follow-up data at both timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU)
Number analyzed (Participants) | 14 | 14 | 14
units on a scale
  12 weeks Mental Health Composite Score | 7.03 (9.94) | 1.51 (8.39) | 5.19 (5.73)
  12 weeks Physical Health Composite Score | 1.88 (9.22) | 0.42 (7.18) | 0.83 (10.61)
  24 weeks Mental Health Composite Score: number analyzed (Participants) | 14 | 13 | 12
  24 weeks Mental Health Composite Score | 7.54 (9.61) | -1.36 (11.32) | 8.28 (8.73)
  24 weeks Physical Health Composite Score: number analyzed (Participants) | 14 | 13 | 12
  24 weeks Physical Health Composite Score | 2.13 (10.07) | 1.00 (8.27) | 0.75 (11.30)

11. Secondary Outcome: Changes in MOS SAS Scores
Description: Three Medical Outcomes Study Specific Adherence Scale (MOS SAS) items assessing medication, diet, and exercise, will be measured individually and as a composite score (Range: 3-18). Change was calculated by subtracting the score at baseline from the score at 12 weeks and 24 weeks. Higher scores indicate better adherence to health behaviors.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: Not all participants provided follow-up data at both timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU)
Number analyzed (Participants) | 14 | 14 | 14
units on a scale
  12 weeks | 2.50 (2.59) | 2.64 (2.27) | 1.14 (2.38)
  24 weeks: number analyzed (Participants) | 14 | 13 | 12
  24 weeks | 2.29 (2.81) | 2.23 (3.56) | 1.42 (1.73)

12. Secondary Outcome: Changes in Sodium Intake (as Measured With the SSQ)
Description: The Scored Sodium Questionnaire (SSQ) is a self-report scale that assesses the frequency with which participants consume a variety of sodium-containing foods, ranging from "Rarely or Never Eaten" to "At Least Once Daily." It is used to calculate daily sodium intake (Range: 0-215). Change was calculated by subtracting the score at baseline from the score at 12 weeks and 24 weeks. Higher scores indicate higher sodium intake.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: Not all participants provided follow-up data at both timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU)
Number analyzed (Participants) | 14 | 14 | 14
units on a scale
  12 weeks | -18.25 (17.62) | -12.93 (15.90) | -11.68 (19.77)
  24 weeks: number analyzed (Participants) | 14 | 13 | 12
  24 weeks | -13.18 (20.14) | -14.65 (20.26) | -0.63 (23.95)

13. Secondary Outcome: Changes in Self-Reported Medication Adherence (SRMA)
Description: The Self-Reported Medication Adherence (SRMA) asks what percent of the time (in 10% increments) participants took all of their medications as prescribed in the past week and in the past 2 weeks (Range: 0-100). Change was calculated by subtracting the score at baseline from the score at 10 weeks.
Time Frame: Baseline, 12 weeks and 24 weeks
Population: Not all participants provided follow-up data at both timepoints.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU)
Number analyzed (Participants) | 14 | 14 | 14
percentage of time
  12 weeks | 43 (51) | 0 (39) | 21 (70)
  24 weeks | 36 (50) | 8 (64) | 8 (100)

14. Secondary Outcome: Change in Physical Activity
Description: Assessed by ActiGraph GT3X+ step counters which are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. We will measure both number of steps per day (primary physical health outcome). Change scores will be calculated by subtracting the number of steps per day at baseline from number of steps per day at 12 weeks and 24 weeks.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: Not all participants provided wore Actigraph GT3X+ step counters or provided follow-up data at both timepoints.
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU)
Number analyzed (Participants) | 12 | 13 | 11
steps/day
  12 weeks: number analyzed (Participants) | 11 | 13 | 11
  12 weeks | 454 (1066) | 409 (1033) | -412 (1305)
  24 weeks: number analyzed (Participants) | 12 | 11 | 10
  24 weeks | 821 (2232) | -330 (1287) | 76 (1207)

15. Secondary Outcome: Change in Moderate to Vigorous Physical Activity
Description: Assessed with ActiGraph GT3X+ step counters, which are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. Change was calculated by subtracting the MVPA at baseline from the MVPA at 12 weeks and 24 weeks.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: Not all participants provided wore Actigraph GT3X+ step counters or provided follow-up data at both timepoints.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU)
Number analyzed (Participants) | 12 | 13 | 11
minutes/day
  12 weeks | 5.72 (10.58) | 0.27 (2.85) | -4.11 (19.02)
  24 weeks | 5.18 (15.02) | -2.66 (4.48) | -1.32 (6.23)

16. Secondary Outcome: Feasibility of Actigraph
Description: Feasibility will be measured by examining the number of participants who provide adequate Actigraph data, defined in this study as at least 480 minutes for 5 days, at each time point.
Time Frame: Baseline, 12 weeks and 24 weeks
Population: Not all participants provided wore Actigraph GT3X+ step counters or provided follow-up data at both timepoints.
Measure: Number; unit: Participants with adequate activity data
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU)
Number analyzed (Participants) | 15 | 15 | 15
Participants with adequate activity data
  12 weeks | 11 | 13 | 11
  24 weeks | 12 | 11 | 10

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from each participant for 6 months, the entire duration of time when they were active in the study.
Arm/Group | PP-based Health Behavior Intervention | MI-based Educational Control Condition | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/15 | 1/15
Other Adverse Events (participants affected / at risk) | 3/15 | 5/15 | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PP-based Health Behavior Intervention (N=15) | MI-based Educational Control Condition (N=15) | Treatment as Usual (TAU) (N=15)
Flu and pneumonia (General disorders) | 0 (0) | 0 (0) | 1 (1) — Participant was hospitalized as a result of having the flu and pneumonia.
Altered mental state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Participant was admitted to the hospital as a result of having an altered mental state.
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Participant was admitted to the hospital after being found to have a urinary tract infection.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PP-based Health Behavior Intervention (N=15) | MI-based Educational Control Condition (N=15) | Treatment as Usual (TAU) (N=15)
Unexpected Shortness of Breath and Weight Gain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Participant reported worsening shortness of breath and weight gain.
Unexpected Chest Pain (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) — 3 participants each reported experiencing chest pain.
Unexpected Shortness of Breath (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Participant reported experiencing shortness of breath.
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Participant went to the ED for a urinary tract infection but was not admitted.
Unexpected Arm Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) — Participant reported experiencing arm pain and thought it was likely attributable to weight lifting exercises.
Fractured foot and ankle (General disorders) | 0 (0) | 1 (1) | 0 (0) — Participant was in a car accident which left them with a fractured foot and ankle.
Unexpected Fall (General disorders) | 0 (0) | 1 (1) | 0 (0) — Participant reported that they had tripped and fell in their home, but that there was no head trauma or need for medical care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT03220204/Prot_SAP_000.pdf